CLINICAL TRIAL: NCT02613117
Title: Research on Oral Tolerability and Product Application/Response of Two Oxalate Products for Dental Patients With Risk of Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014067
Record Dates: First submitted 2015-11-13; First posted 2015-11-24 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Dentinal Hypersensitivity

ARMS (2):
- potassium oxalate gel (Other): potassium oxalate gel self applied
  Interventions: Device: Potassium Oxalate Gel
- oxalate liquid, SnF2 paste (Other): Potassium oxalate liquid professionally applied, Stannous fluoride paste self applied
  Interventions: Device: Potassium Oxalate Liquid; Drug: Stannous fluoride paste

INTERVENTIONS:
Device: Potassium Oxalate Gel — Self applied
  Arms: potassium oxalate gel
Device: Potassium Oxalate Liquid — Professionally Applied
  Arms: oxalate liquid, SnF2 paste
Drug: Stannous fluoride paste — SnF2 Paste
  Arms: oxalate liquid, SnF2 paste

SUMMARY:
This study will assess the oral tolerability and immediate post-treatment safety of topical application for two marketed oxalate products as initial care in dental patients to treat or prevent tooth sensitivity pain that may be attributed to dentinal hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* sign an informed consent form and be given a copy
* be in good general health as determined by the Investigator/designee
* agree to not participate in any other oral care study for the duration of this study
* agree to return for scheduled visits and follow all study procedures
* have at least one tooth at risk for hypersensitivity.

Exclusion Criteria:

* any medical condition requiring pre-medication prior to dental procedures
* any diseases or conditions that might interfere with the subject safely completing the study
* inability to undergo study procedures
* a history of kidney stones
* have self-reported pregnancy or nursing
* known allergies to the following ingredients; aqua, glycerin, cellulose gum, dipotassium oxalate, carbomer, sodium hydroxide, sodium benzoate, or potassium sorbate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Potassium Oxalate Gel | Oxalate Liquid, SnF2 Paste
Started | 57 | 47
Completed | 57 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Potassium Oxalate Gel | Oxalate Liquid, SnF2 Paste | Total
Number analyzed (Participants) | 57 | 47 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (11.99) | 45.8 (12.91) | 43.6 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 35 | 76
  Male | 16 | 12 | 28
Region of Enrollment [Number; unit: participants]
  United States | 57 | 47 | 104

OUTCOME MEASURES:

1. Primary Outcome: How Satisfied Were Participants With Treatment?
Description: Questionnaire indicating the frequencies of using various oral hygiene products by subjects at 5 different dental practices.
Time Frame: up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Potassium Oxalate Gel | Oxalate Liquid, SnF2 Paste
Number analyzed (Participants) | 56 | 44
Participants
  Very Dissatisfied | 0 | 1
  Somewhat Dissatisfied | 2 | 2
  Neutral | 7 | 11
  Somewhat Satisfied | 23 | 10
  Very Satisfied | 24 | 20

2. Primary Outcome: Ease of Treatment at Home
Description: as for outcome 1
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Potassium Oxalate Gel | Oxalate Liquid, SnF2 Paste
Number analyzed (Participants) | 56 | 44
Participants
  Extremely Difficult to Use | 0 | 0
  Somewhat Difficult to Use | 1 | 0
  Neither Easy Nor Difficult to Use | 2 | 12
  Somewhat Easy to Use | 24 | 2
  Extremely Easy to Use | 29 | 30

3. Primary Outcome: Did Participants Notice a Difference in the Areas Noted?
Description: as for outcome 1
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Potassium Oxalate Gel | Oxalate Liquid, SnF2 Paste
Number analyzed (Participants) | 56 | 44
Participants
  Hot/Cold: Yes | 42 | 30
  Hot/Cold: No | 14 | 14
  Sweet/Sour: Yes | 19 | 9
  Sweet/Sour: No | 37 | 35
  Hard/Soft: Yes | 7 | 13
  Hard/Soft: No | 49 | 31
  Cold Air: Yes | 28 | 18
  Cold Air: No | 28 | 26
  Other: Yes | 8 | 9
  Other: No | 48 | 35

ADVERSE EVENTS:
Arm/Group | Potassium Oxalate Gel | Oxalate Liquid, SnF2 Paste
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/47
Other Adverse Events (participants affected / at risk) | 0/57 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI should disclose plans to sponsor prior to public release.